CLINICAL TRIAL: NCT03904472
Title: Single-arm Pilot Trial of Web-based Cognitive Behavioral Therapy for Insomnia (CBTI) in Gastroesophageal Reflux Disease (GERD) Patients With Insomnia
Brief Title: Cognitive Behavioral Therapy for Insomnia (CBTI) in GERD Patients With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Gastroenterological Association (Other)
Responsible Party: Principal Investigator, Joan Chen, Clinical Assistant Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00157452
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2021-06

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: cognitive behavioral therapy; GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-based CBTI (Experimental): Participants will have 8 weeks to receive 6 therapy sessions. Content is dynamically driven by an animated therapist who guides the user through the program.
  Interventions: Behavioral: Web-based CBTI

INTERVENTIONS:
Behavioral: Web-based CBTI — Sessions comprise a range of cognitive and behavioral techniques and psychoeducation including sleep hygiene. During the intervention period the participant will complete daily online sleep diaries. Additionally, participants will be asked to complete multiple questionnaires.

SUMMARY:
This study will enroll patients with persistent reflux symptoms despite proton-pump inhibitor therapy and chronic insomnia. Participants that are eligible for the study and agree to participate will receive cognitive behavioral therapy for insomnia (CBTI) delivered by a web-based approach. The goal of the treatment is to improve the participants insomnia and reflux symptoms. In addition to the cognitive behavioral therapy, participants will be asked to keep a daily diary and periodically complete questionnaires to assess their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent reflux symptoms (GERDQ >8) despite proton-pump inhibitor (PPI) therapy.
* Patients screened positive for chronic insomnia (insomnia severity index [ISI] ≥15).

Exclusion Criteria:

* Patients with major esophageal motility disorder, prior foregut surgeries, severe cardiopulmonary diseases, or major psychological comorbidities.
* Patients who report being in "poor" or "very poor" physical or mental health.
* Patients with sleep apnea (based on STOP-BANG questionnaire >4)
* Patients with AUDIT score >15, indicating alcohol dependence
* Patients regularly taking medications for sleep >2 times per week who cannot stop the sleep aid at least 4 weeks prior to and during the study trial.
* Patients who have previously undergone CBT for insomnia (in person or online).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Reflux Symptom Questionnaire-7-day recall (RESQ-7) | up to 8 weeks post treatment
  RESQ-7 contains 13 items which are aggregated to 4 frequency and 4 intensity domain scores: heartburn (5 items), regurgitation (4 items), cough, hoarseness, difficulty swallowing (3 items), burping (1 item).
  Frequency questions are scored from 0-7 and intensity questions are scored from 0-5. The range of scores are 0-156 (0 meaning no symptoms, 156 being the worst).
Gastroesophageal Reflux Disease Quality of Life (GERD-QoL) | up to 8 weeks post treatment
  The questionnaire is composed of 6 items, 4 of which assess symptoms and situations considered positive predictors for GERD diagnosis: heartburn, regurgitations, disorders related to sleep and use of over the counter products. Other 2 items assess 2 nausea and epigastric pain. Participants answer each question about symptoms frequency during last week using a Likert like scale from 0 to 3 for positive predictors and from 3 to 0 for negative predictors. The maximum score that can be obtained is 18.

SECONDARY OUTCOMES:
Insomnia severity index (ISI) | up to 8 weeks post treatment
  ISI is a 7-item psychometrically validated measure used to rate insomnia.The total score ranges from 0-28 where higher values indicate increased severity of insomnia.
Sleep Onset Latency (SOL) | up to 8 weeks post treatment
  This is based on the participants sleep diary and how many minutes it took the participants to fall asleep.
Wake After Sleep Onset (WASO) | up to 8 weeks post treatment
  This is based on the participants sleep diary and how many minutes they woke up after sleeping.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Chen, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan GI Physiology Lab, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No